CLINICAL TRIAL: NCT02402439
Title: Treatment of Type I Diabetes by Islet Transplantation Into the Gastric Submucosa Study Protocol
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Andrew Posselt (Other)
Responsible Party: Sponsor-Investigator, Andrew Posselt, Professor of Surgery in Residence, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IGS
Record Dates: First submitted 2015-03-18; First posted 2015-03-30 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 diabetes; diabetes mellitus; pancreatic islet transplant; beta cell replacement
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Pancreatic Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Islet Transplant (Experimental): Islet transplantation into the gastrointestinal submucosa
  Interventions: Drug: Islet cells; Procedure: Islet transplantation into the gastrointestinal submucosa

INTERVENTIONS:
Drug: Islet cells — Transplantation of islets into the gastrointestinal submucosa
  Other Names: pancreas
Procedure: Islet transplantation into the gastrointestinal submucosa — Transplantation of islets into the gastrointestinal submucosa
  Other Names: pancreas

SUMMARY:
The goal of this trial is to gain initial clinical experience regarding the safety and efficacy of treating type I diabetes in people who have received a kidney transplant by transplanting islets into a new transplant site in the stomach (gastrointestinal submucosa). A total of 6 patients will be enrolled in the study and followed for a period of up to 3 years after the last islet transplant.

DETAILED DESCRIPTION:
Pancreatic islet transplantation offers a minimally invasive approach to restore normoglycemia in type 1 diabetics while avoiding the hypoglycemic complications observed with intensive insulin therapy and the surgical complications associated with pancreas transplantation. Although significant progress has been made in clinical islet transplantation, overall outcomes remain suboptimal since many patients lose insulin independence a few years after transplantation and multiple donors are usually needed to achieve independence. The cause of this progressive loss of function is multifactorial, but mounting evidence suggests that much of the islet loss after transplant is directly related to the intraportal transplant site that is used in clinical islet transplantation. Intravascular infusion of the islets triggers a severe,non-specific inflammatory response (immediate blood-mediated inflammatory reaction, IBMIR) which destroys at least 50% of the islet mass. The engraftment of the surviving islets is further compromised by the relatively hypoxic portal venous environment, and the infused islets are exposed to potentially toxic levels of immunosuppressive agents being absorbed from the gut into the portal circulation. Together, these characteristics contribute to early as well as late loss of islet function after transplantation. The gastrointestinal submucosa is a newly described transplant site that can support islet engraftment while avoiding many of the drawbacks associated with intraportal infusion. In addition, this site is easily accessible via upper endoscopy and the submucosal injection procedure is safe and technically straightforward.

The aim of this prospective, single-center trial is to provide initial clinical experience regarding the safety and efficacy of endoscopic gastric and duodenal submucosal islet transplantation in type I diabetic patients with kidney allografts. A total of 6 patients will be recruited into the trial. The investigators will follow the standardized islet manufacturing protocols and the thymoglobulin-based induction immunosuppressive regimen developed by the Clinical Islet Transplant consortium (CIT). Outcomes will include safety measures, glycemic control and insulin use, metabolic assessments of graft function, allo/auto-immune responses, and protocol biopsies to assess graft rejection/inflammation. The investigators believe that this novel approach to islet transplantation has the potential to significantly improve current islet transplantation outcomes by enhancing islet engraftment and long-term function.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects age 18 to 70 years of age.
2. Subjects who are able to provide written informed consent and to comply with study procedures.
3. Clinical history compatible with T1D (onset < 40 yrs old and insulin dependent for > 5 yrs at enrollment.
4. Absent stimulated c-peptide (< 0.3 ng/mL) in response to a (Boost® 6 mL/kg BW to a maximum of 360 mL; another equivalent product), measured at 60 and 90 min after start of consumption.
5. Subjects who are > 3 months post-renal transplant who are taking appropriate calcineurin inhibitor (CNI) based maintenance immunosuppression ([tacrolimus alone or in conjunction with sirolimus, mycophenolate mofetil, myfortic, or azathioprine; or cyclosporine in conjunction with sirolimus, mycophenolate mofetil, or myfortic ± Prednisone ≤ 10 mg/day).
6. Stable renal function as defined by a creatinine of no more than one third greater than the average creatinine determination performed in the 3 previous months prior to islet transplant, until rejection, obstruction or infection is ruled out.
7. Reduced awareness of hypoglycemia manifested a Clarke score >4 and at least 1 episode of severe hypoglycemia in the past 12 months prior to study enrollment. This criterion requires that there has been involvement in intensive diabetes management under the direction of an endocrinologist, diabetologist, or diabetes specialist prior to study enrollment. Intensive diabetes management is defined as self-monitoring of glucose values no less than 3 times each day averaged over each week and by the administration of three or more insulin injections each day or insulin pump therapy. Severe hypoglycemia is defined as an event with one of the following symptoms: memory loss; confusion; uncontrollable behavior; irrational behavior; unusual difficulty in awakening; suspected seizure; seizure; loss of consciousness; or visual symptoms, and which was associated with either a BG level < 54 mg/dl [3.0 mmol/L] or prompt recovery after oral carbohydrate, IV glucose, or glucagon administration.

Exclusion Criteria:

1. Weight more than 100 kg or body mass index (BMI) > 30 kg/m2.
2. Insulin requirement of >1.0 IU/kg/day or <15 U/day.
3. Other (non-kidney) organ transplants except prior failed pancreatic graft where graft failure is attributed to thrombosis within the first 4 weeks or to other technical reasons that require graft pancreatectomy; with the graft pancreatectomy occurring more than 6 months prior to enrollment.
4. Untreated or unstable proliferative diabetic retinopathy.
5. Blood Pressure: SBP > 160 mmHg or DBP >100 mmHg despite treatment with antihypertensive agents.
6. Calculated GFR of ≤ 40 mL/min/1.73 m2 using the subject's measured serum creatinine and the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation. (59)
7. Proteinuria (albumin/creatinine ratio or ACr > 300mg/g) of new onset since kidney transplantation.
8. Calculated panel-reactive anti-HLA antibodies > 50%. Subjects with calculated panel reactive anti-HLA antibodies ≤ 50% will be excluded if any of the following are detected:

   * Positive cross-match
   * Islet donor-directed anti-HLA antibodies detected by Luminex® Single Antigen/specificity bead assay including weakly reactive antibodies that would not be detected by a flow cross-match
9. For female subjects: Positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of the study and 4 months after discontinuation. For male subjects: intent to procreate during the duration of the study or within 4 months after discontinuation or unwillingness to use effective measures of contraception. Oral contraceptives, Norplant®, Depo-Provera®, and barrier devices with spermicide are acceptable contraceptive methods; condoms used alone are not acceptable.
10. Active infection including hepatitis B, hepatitis C, HIV, or TB. A positive skin test (PPD) in itself is not an exclusion, and will be followed up by a QuantiFERON® gold assay.
11. Negative screen for EBV IgG.
12. Invasive Aspergillus, Histoplasmosis, and Coccidioidomycosis infection within 1 year prior to study entry.
13. Any history of malignancy except for completely resected squamous or basal cell carcinoma of the skin.
14. Known active alcohol or substance abuse.
15. Severe co-existing cardiac disease, characterized by any one of these conditions:

    * Recent MI (within past 6 months),
    * Evidence of ischemia on functional cardiac exam within the last year,
    * Left ventricular ejection fraction < 30%,
    * Valvular disease requiring replacement with prosthetic valve.
16. Persistent elevation of liver function tests at time of study entry. Persistent SGOT (AST), SGPT (ALT), alkaline phosphatase values > 1.5, or total bilirubin > 1 times normal upper limits will exclude a subject.
17. Active infections (except mild skin and nail fungal infections).
18. Acute or chronic pancreatitis.
19. Active peptic ulcer disease or gastritis, symptomatic gallstones, or portal hypertension.
20. Treatment with any anti-diabetic medication other than insulin within 4 weeks of enrollment.
21. Use of any investigational agents within 4 weeks of enrollment.
22. Administration of live attenuated vaccine(s) within 2 months of enrollment.
23. Any medical condition that, in the opinion of the investigator, will interfere with safe study completion.
24. Positive screen for BK viremia at time of screening.
25. Untreated hyperlipidemia - TC > 200 mg/dL, TGC > 200 mg/dL, LDL > 130 mg/dL
26. Use of glucocorticoids for non-transplant-related indications.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Insulin independence | 75 days after the first transplant
  off insulin therapy for at least 1 week and all of the following criteria are met:
  * HbA1c < 6.5% or a > 2.5% decrease from baseline;
  * Daily fasting capillary glucose should not exceed 140 mg/dL (7.8 mmol/L) more than 3 times in the past week;
  * 2-hour post-prandial capillary glucose should not exceed 180 mg/dl (10.0 mmol/L) more than three times in the past week;
  * Fasting plasma glucose < 126 mg/dL (7.0 mmol/L); if the fasting plasma glucose is > 126 mg/dL (7.0 mmol/L), it must be confirmed in an additional one out of two measurements; Protocol Version 4.0 December 19, 2017 39
  * Evidence of endogenous insulin production defined as fasting or stimulated C-peptide >0.5 ng/mL (0.16 nmol/L).
Insulin independence | 1 year after the first transplant
  off insulin therapy for at least 1 week and all of the following criteria are met:
  * HbA1c < 6.5% or a > 2.5% decrease from baseline;
  * Daily fasting capillary glucose should not exceed 140 mg/dL (7.8 mmol/L) more than 3 times in the past week;
  * 2-hour post-prandial capillary glucose should not exceed 180 mg/dl (10.0 mmol/L) more than three times in the past week;
  * Fasting plasma glucose < 126 mg/dL (7.0 mmol/L); if the fasting plasma glucose is > 126 mg/dL (7.0 mmol/L), it must be confirmed in an additional one out of two measurements; Protocol Version 4.0 December 19, 2017 39
  * Evidence of endogenous insulin production defined as fasting or stimulated C-peptide >0.5 ng/mL (0.16 nmol/L).
Insulin independence | 1 year after the last transplant
  off insulin therapy for at least 1 week and all of the following criteria are met:
  * HbA1c < 6.5% or a > 2.5% decrease from baseline;
  * Daily fasting capillary glucose should not exceed 140 mg/dL (7.8 mmol/L) more than 3 times in the past week;
  * 2-hour post-prandial capillary glucose should not exceed 180 mg/dl (10.0 mmol/L) more than three times in the past week;
  * Fasting plasma glucose < 126 mg/dL (7.0 mmol/L); if the fasting plasma glucose is > 126 mg/dL (7.0 mmol/L), it must be confirmed in an additional one out of two measurements; Protocol Version 4.0 December 19, 2017 39
  * Evidence of endogenous insulin production defined as fasting or stimulated C-peptide >0.5 ng/mL (0.16 nmol/L).

SECONDARY OUTCOMES:
Changes in HbA1c | From day 28 to 365
  Proportion of subjects with an HbA1c <7.0% and free of severe hypoglycemic events from day 28 to 365 after the first and final islet transplant
Changes (reduction) in insulin requirements | up to 5 years
  decrease of insulin dose as compared to pre-transplantation of islets
Incidence of adverse events | up to 5 years
  the incidence of AEs related to the transplant procedure or immunosuppression

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Posselt, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No